CLINICAL TRIAL: NCT04345471
Title: A Placebo-controlled Study of MD-120 in Patients With Depression
Brief Title: A Study of MD-120 in Patients With Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD120101; JapicCTI-205252 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2020-04-06; First posted 2020-04-14 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MD-120 100 mg (Experimental)
  Interventions: Drug: Desvenlafaxine 100 mg
- MD-120 50 mg (Experimental)
  Interventions: Drug: Desvenlafaxine 50 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine 100 mg — once daily dosing for 8 weeks
  Arms: MD-120 100 mg
Drug: Desvenlafaxine 50 mg — once daily dosing for 8 weeks
  Arms: MD-120 50 mg
Drug: Placebo — once daily dosing for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to verify the efficacy and evaluate the safety of 8-week once-daily oral administration of MD-120 in Japanese patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of Major Depressive Disorder (MDD) based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5).
* Hamilton Depression Rating Scale-17 (HAM-D17) total score of ≥20.

Exclusion Criteria:

* Patient who meets DSM-5 criteria of the following disorders for current or past history.

Schizophrenia spectrum and other psychotic disorders Bipolar and related disorders Substance use disorders (exclusive of tobacco and caffeine)

* Patient who had suicidal behavior in Columbia-Suicide Severity Rating Scale (C-SSRS) within 1 year before start of screening phase.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Hayashi, Study Director — Mochida Pharmaceutical Company, Ltd.
Locations (1):
- Mochida Investigational sites, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 82 investigational sites in Japan from 18 May 2020 to 14 September 2022.
Pre-assignment Details: Participants who met entry criteria were enrolled placebo lead-in period for one week prior to randomization, after that participants randomized and enrolled in one of three treatment group (Placebo group, MD-120 50 mg group, MD-120 100 mg group) for 8 weeks as double-blind treatment period.
Groups:
- Placebo: Placebo, orally, once daily for up to Week 8
- MD-120 50 mg: MD-120 50 mg, orally, once daily for up to Week 8
- MD-120 100 mg: MD-120 50 mg, orally, once daily for up to Week 1, followed by MD-120 100 mg, orally, once daily for up to Week 8
Period: Overall Study
Arm/Group | Placebo | MD-120 50 mg | MD-120 100 mg
Started | 204 | 207 | 204
Received Treatment | 204 | 206 | 204
Completed | 185 | 195 | 186
Not Completed | 19 | 12 | 18
Not completed — Adverse Event | 8 | 5 | 6
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Withdrawal by Subject | 10 | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MD-120 50 mg | MD-120 100 mg | Total
Number analyzed (Participants) | 203 | 206 | 204 | 613
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (12.0) | 39.8 (12.1) | 39.6 (12.7) | 39.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 104 | 91 | 297
  Male | 101 | 102 | 113 | 316
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 203 | 206 | 204 | 613
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 203 | 206 | 204 | 613
Montgomery Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: Scores on a scale] | 31.6 (4.9) | 32.0 (4.7) | 31.5 (4.7) | 31.7 (4.8)
Hamilton Depression Rating Scale-17 (HAM-D17) Total Score [Mean (Standard Deviation); unit: Scores on a scale] | 24.3 (2.9) | 24.3 (3.0) | 23.8 (2.8) | 24.1 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Total MADRS Score From the Baseline to Week 8 Visit During the Treatment Period
Description: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score: Scale ranges from 0 to 60 with a higher score indicating worsening symptoms of depression. Estimates were based on a Mixed-effects Model for Repeated Measures (MMRM) model with the treatment group, assessment timepoint, and the interaction between the treatment group and assessment timepoint as a factor and total MADRS score at baseline as a covariate.
Time Frame: 8 weeks
Population: Of subjects registered for randomization, those meeting all the following items were included in the full analysis set (FAS).
  1. Subjects who received the investigational drug at least once during the treatment period.
  2. Subjects who were evaluated for the total MADRS score at the baseline and at least one timepoint after the start of the treatment period.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | MD-120 50 mg | MD-120 100 mg
Number analyzed (Participants) | 203 | 206 | 204
Score on a scale | -10.4 (0.7) | -11.1 (0.7) | -11.9 (0.7)
Statistical Analysis 1: Comparison: Placebo vs MD-120 50 mg; Test type: Superiority — To adjust for the multiplicity, only when the superiority of MD-120 50 mg to Placebo was verified, the superiority of MD-120 100 mg to Placebo was tested; p = 0.509, MMRM — A priori threshold for statistical significance is p<0.05, 2-sided; LS mean difference = -0.6, 95% CI 2-sided [-2.5 to 1.2]
Statistical Analysis 2: Comparison: Placebo vs MD-120 100 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.131, MMRM — A priori threshold for statistical significance is p<0.05, 2-sided. The value was based on the post-hoc analysis by not taking into account the multiplicity; LS mean difference = -1.4, 95% CI 2-sided [-3.3 to 0.4]

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any undesirable or unintended sign (including abnormal findings in general laboratory tests, body weight, and standard 12-lead ECG), symptom, or disease in a subject given the investigational drug, irrespective of the causal relationship to the investigational drug.
Time Frame: 10 weeks
Population: Of subjects registered for randomization, those meeting all the following items will be included in the safety analysis set in treatment period.
  1. Subjects who have received the investigational drug at least once during the treatment period.
  2. Subjects in whom the safety evaluation data after the dose of the investigational drug in the treatment period are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MD-120 50 mg | MD-120 100 mg
Number analyzed (Participants) | 204 | 206 | 204
Participants | 102 | 117 | 124

3. Secondary Outcome: Changes in Total HAM-D17 Score From the Baseline to Week 8 Visit During the Treatment Period
Description: Hamilton Depression Rating Scale-17 (HAM-D17) Total Score: Scale ranges from 0 to 52 with a higher score indicating worsening symptoms of depression. Estimates were based on a MMRM model with the treatment group, assessment timepoint, and the interaction between the treatment group and assessment timepoint as a factor and total HAM-D17 score at baseline as a covariate.
Time Frame: 8 weeks
Population: Of subjects registered for randomization, those meeting all the following items were included in the FAS.
  1. Subjects who received the investigational drug at least once during the treatment period.
  2. Subjects who were evaluated for the total MADRS score at the baseline and at least one timepoint after the start of the treatment period.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | MD-120 50 mg | MD-120 100 mg
Number analyzed (Participants) | 203 | 206 | 204
Scores on a scale | -8.3 (0.5) | -8.4 (0.5) | -8.8 (0.5)
Statistical Analysis 1: Comparison: Placebo vs MD-120 50 mg; Test type: Superiority; p = 0.811, MMRM — A priori threshold for statistical significance is p<0.05, 2-sided; LS mean difference = -0.2, 95% CI 2-sided [-1.5 to 1.2]
Statistical Analysis 2: Comparison: Placebo vs MD-120 100 mg; Test type: Superiority; p = 0.424, MMRM — A priori threshold for statistical significance is p<0.05, 2-sided; LS mean difference = -0.5, 95% CI 2-sided [-1.9 to 0.8]

4. Secondary Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Time Frame: 10 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Plasma Concentration of Desvenlafaxine
Time Frame: Week 2 through week 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebo | MD-120 50 mg | MD-120 100 mg
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/206 | 0/204
Serious Adverse Events (participants affected / at risk) | 2/204 | 3/206 | 2/204
Other Adverse Events (participants affected / at risk) | 43/204 | 67/206 | 71/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=204) | MD-120 50 mg (N=206) | MD-120 100 mg (N=204)
COVID-19 (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=204) | MD-120 50 mg (N=206) | MD-120 100 mg (N=204)
Nausea (Gastrointestinal disorders) | 14 | 27 | 35
Somnolence (Nervous system disorders) | 7 | 13 | 18
Dizziness (Nervous system disorders) | 2 | 16 | 15
Weight decreased (Investigations) | 1 | 5 | 12
Pyrexia (General disorders) | 11 | 10 | 8
Nasopharyngitis (Infections and infestations) | 13 | 9 | 8
Headache (Nervous system disorders) | 3 | 15 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the Study results at any time without the prior written approval of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04345471/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT04345471/SAP_001.pdf